CLINICAL TRIAL: NCT06625593
Title: A Phase 1a/b, Open-label, Multicenter Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of BG-C137, an Antibody-Drug Conjugate Targeting FGFR2b, in Patients With Advanced Solid Tumors
Brief Title: A First-in-Human (FIH) Study of BG-C137, an Anti-Fibroblast Growth Factor Receptor 2b (FGFR2b) Antibody Drug Conjugate, in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BG-C137-101; 2025-523572-23-00 (EU CTIS Number); CTR20244835 (Other: ChinaTrialDrugs)
Record Dates: First submitted 2024-09-23; First posted 2024-10-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor
Keywords: BG-C137; Advanced Solid Tumor; First-in-human; FGFR2b; ADC; Fibroblast growth factor receptor 2b
MeSH Terms: interventions — Antineoplastic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1a: Monotherapy Dose Escalation and Safety Expansion (Experimental): Sequential cohorts of increasing dose levels of BG-C137 will be evaluated as monotherapy
  Interventions: Drug: BG-C137
- Phase 1a: Combination Therapy Dose Confirmation and Safety Expansion (Experimental): Sequential cohorts will be evaluated to confirm the safety levels of BG-C137 in combination with other anticancer agents at selected dose levels that have been determined to be safe in Monotherapy Dose Escalation
  Interventions: Drug: BG-C137; Drug: Anticancer Agents
- Phase 1b: Dose Expansion (Experimental): Recommended Dose(s) of BG-C137 as determined from Ph1a will be evaluated in select indications
  Interventions: Drug: BG-C137

INTERVENTIONS:
Drug: BG-C137 — Administered intravenously
Drug: Anticancer Agents — Administered intravenously or orally
  Arms: Phase 1a: Combination Therapy Dose Confirmation and Safety Expansion

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary antitumor activity of BG-C137 alone and in combination with anticancer agents in participants with advanced solid tumors. The study will be conducted in two phases: Phase 1a (Monotherapy Dose Escalation, and Safety Expansion; Combination Dose Confirmation and Safety Expansion) and Phase 1b (Dose Expansion).

DETAILED DESCRIPTION:
Our company, previously known as BeiGene, is now officially BeOne Medicines. Because some of our older studies were sponsored under the name BeiGene, you may see both names used for this study on this website.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced or metastatic solid tumors.
2. Life expectancy of ≥ 3 months.
3. Prior standard systemic therapy in the advanced or metastatic setting. Dose Escalation: Participants for whom further standard treatment is not available, not tolerated or determined not appropriate based on the investigator's judgment. Combo Dose Confirmation, Combo Safety Expansion, and Dose Expansion: Participants who have received at least 1 or 2 prior lines of systemic therapy, which included a fluoropyrimidine and/or a platinum in the advanced or metastatic setting
4. Tumors with FGFR2b expression/ or FGFR2 gene amplification. Participants must provide agreement for collection of archival tissue or recently obtained fresh tumor biopsy for central evaluation of FGFR2b expression levels and other biomarker assessments.
5. ≥ 1 measurable lesion per RECIST v1.1.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
7. Adequate organ function as determined per protocol.

Exclusion Criteria:

1. Prior exposure to topoisomerase I inhibitor (TOP1i)-based antibody-drug conjugate (ADC) therapies or FGFR2b-targeted ADC therapies.
2. Active or chronic corneal disorder, history of corneal transplantation, corneal keratitis, keratoconjunctivitis, keratopathy, corneal abrasion, inflammation or ulceration, other active ocular conditions and any clinically significant corneal disease that prevents adequate monitoring of drug-induced keratopathy.
3. Spinal cord compression, or active leptomeningeal disease or uncontrolled, untreated brain metastasis.
4. Systemic antitumor therapy (including targeted therapy and immunotherapy ≤ 14 days, ≤ 28 days for immuno- oncological antibody, ≤ 14 days or 5 half-lives [whichever is shorter] for chemotherapy, ADCs, or investigational therapy) before first dose of study drug(s).
5. Toxicities due to prior therapy that have not recovered.
6. Any malignancy ≤ 2 years before first dose of study drug(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively.
7. History of interstitial lung disease (ILD), noninfectious pneumonitis, oxygen saturation at rest < 92%, or requirement for supplemental oxygen at baseline.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 2 years
  Number of participants with AEs and SAEs as graded by the National Cancer Institute- Common Terminology Criteria for Adverse Events Version (NCI CTCAE 5.0)), including AEs that meet protocol-defined dose-limiting toxicity (DLT) criteria and AEs meeting protocol-defined adverse event of clinical interest (AECIs)
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of BG-C137 | Up to approximately 2 years
  The MTD or MAD is defined as the highest dose evaluated for which the estimated toxicity rate is closest to a target toxicity rate, or the highest dose administered, respectively.
Phase 1a: Recommended Dose(s) for Expansion (RDFE[s]) of BG-C137 as monotherapy and in combination with anticancer agents | Up to approximately 2 years
  RDFE(s) is determined based on relevant data, as available
Phase 1b: The recommended Phase 2 dose (RP2D) of BG-C137 | Up to approximately 2 years
  The RP2D of BG-C137 monotherapy will be determined based on relevant data, as available
Phase 1b: Overall Response Rate (ORR) | Up to approximately 2 years
  ORR is defined as the percentage of participants with confirmed complete response (CR) or partial response (PR) by Response Evaluations Criteria in Solid Tumors Version 1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Phase 1a: ORR | Up to approximately 2 years
  ORR is defined as the percentage of participants with CR or PR, as determined by RECIST v1.1
Phase 1a and 1b: Disease Control Rate (DCR) | Up to approximately 2 years
  DCR is defined as the percentage of participants with best overall response of a CR, PR, and stable disease, as assessed by RECIST v1.1
Phase 1a and 1b: Duration of Response (DOR) | Up to approximately 2 years
  DOR is defined as the time from the first determination of an objective response per RECIST v1.1 until the first documentation of progression or death, whichever comes first, as assessed using RECIST v1.1
Phase 1b: Progression Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the date of the first dose of study drug to the date of the first documentation of progressive disease assessed using RECIST v1.1 or death, whichever occurs first
Phase 1b: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 2 years
  Number of participants with AEs and SAEs as graded by the National Cancer Institute- Common Terminology Criteria for Adverse Events Version (NCI CTCAE 5.0), and AEs meeting protocol-defined adverse event of clinical interest (AECI)s.
Phase 1a: Plasma concentrations of BG-C137 analytes | Up to approximately 1 year; at the end of treatment (maximum of 2 years) and at the first safety follow-up visit (30 days after last dose)
Phase 1b: Plasma concentrations of BGB-C137 analytes | Up to approximately 1 year; at the end of treatment (maximum of 2 years) and at the first safety follow-up visit (30 days after last dose)
Phase 1a: Maximum observed plasma concentration (Cmax) of BGB-C137 analytes | Twice in the first 3 months
Phase 1a: Time to reach maximum observed plasma concentration (Tmax) of BGB-C137 analytes | Twice in the first 3 months
Phase 1a: Minimum Observed Plasma Concentration (Ctrough) Of BGB-C137 analytes | Twice in the first 3 months
Phase 1a: Area Under the Plasma Concentration-time Curve (AUC) of BGB-C137 analytes | Twice in the first 3 months
Phase 1a: Terminal Half-Life (t1/2) of BGB-C137 analytes | Twice in the first 3 months
Phase 1a and 1b: Incidence of Antidrug Antibodies (ADAs) to BGB-C137 | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (31):
- United States (6):
  - Usc Norris Comprehensive Cancer Center (Nccc), Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Md Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Australia (5):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Icon Cancer Centre South Brisbane, South Brisbane, Queensland
  - Monash Health, Clayton, Victoria
  - Cabrini Hospital Malvern, Malvern East, Victoria
- China (11):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The Tumor Hospital Affiliated to Guangxi Medical Universitywuxiang Branch, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Affiliated Hospital of Jiangnan University South Campus, Wuxi, Jiangsu
  - The Affiliated Hospital of Qingdao University Branch North, Qingdao, Shandong
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital Branch Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
- South Korea (9):
  - Cha Bundang Medical Center, Cha University, BundangGu SeongnamSi, Gyeonggi-do
  - Seoul National University Bundang Hospital, BundangGu SeongnamSi, Gyeonggi-do
  - Kyungpook National University Chilgok Hospital, BukGu, Gyeongsangbukdo
  - Gachon University Gil Medical Center, NamdongGu, Incheon Gwang'yeogsi
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/